CLINICAL TRIAL: NCT07252986
Title: A Multi-omics Breast Cancer Distant Metastasis Prediction Model Empowered by Artificial Intelligence and Its Clinical Translation Research
Brief Title: Clinical Translation Research on a Multi-omics Breast Cancer Distant Metastasis Prediction Model Empowered by Artificial Intelligence
Acronym: COMPASS-BC
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Jian Huang, Head of Breast Surgery Department, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2025-COMPASS-BC; 2025-COMPASS-BC (Other: The Second Affiliated Hospital, Zhejiang University School of Medicine)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Breast; Breast Cancer; Pathology
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Based on the study protocol, the following specific types of biological samples will be collected, processed, and retained:
  * Primary tumor tissue
  * Metastatic tumor tissue, specifically from liver, lung, bone, and brain metastases
  * Paired samples of primary and metastatic tumors (with a goal of over 1,000 pairs)
  * Blood samples, which will be used for liquid biopsy
  * The informed consent form specifies the collection of 6-10ml of peripheral blood
  * Data from previously retained biological samples, such as plasma
  * Patient-derived breast organoids All collected samples will be stored at -80°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Metastatic Risk Stratification (High/Medium/Low Risk)
- Group 2: Organ-Specific Metastasis (Bone/Lung/Liver/Brain)
- Group 3: Non-Metastatic Control Group

SUMMARY:
Breast cancer is one of the most common malignancies in women worldwide, and distant metastasis is the main cause of poor prognosis and death. This project aims to construct a precision prediction system based on multi-omics (digital pathology, immunohistochemistry, proteomics, gene sequencing) and artificial intelligence to predict distant and organ-specific metastasis (bone, lung, liver, brain) in breast cancer, analyze its mechanisms, and provide new solutions for precision medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients pathologically diagnosed with breast cancer at our hospital or participating centers between January 1, 2000, and December 30, 2028.
2. Must meet one of the following: 1) Initially diagnosed with breast cancer at our hospital, has developed distant metastasis (liver, bone, lung, or brain), and has a biopsy or surgical specimen from the metastatic site stored at our hospital, with complete clinical information available. 2) Primary tumor specimen is not at our hospital, but a biopsy or surgical specimen from a distant metastatic site (liver, bone, lung, brain) is stored at our hospital.

Exclusion Criteria:

1. Concomitant metastatic malignancy from another primary cancer.
2. Incomplete clinical information.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises female patients diagnosed with breast cancer between 2000 and 2028, identified through participating hospital centers. This includes patients who have developed distant (organ-specific) metastasis (liver, lung, bone, or brain) and for whom primary and/or metastatic tissue samples are available.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Metastasis-Free Survival | From diagnosis up to December 30, 2028
  Time from initial breast cancer diagnosis to the occurrence of distant metastasis.

SECONDARY OUTCOMES:
Performance of Prediction Models | At the end of the study (December 2028)
  Evaluate the performance of (1) the metastatic risk stratification model, (2) the organ-specific metastasis prediction model, and (3) the metastasis time-window prediction model.
  Measure: Accuracy and Area Under the Curve (AUC). (Target accuracy ≥80%, AUC ≥0.80)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is not guaranteed and is strictly conditional. First, consent for the long-term storage and future research use of data is collected as a separate, optional item on the Informed Consent Form. Therefore, IPD cannot be shared from any participant who does not provide this specific optional consent.
  Second, the study involves highly sensitive multi-modal data, including digital pathology, proteomics, and genomic sequencing. This data is subject to strict privacy-preserving protocols (such as encryption and differential privacy) and oversight by the institutional data security committee to protect participant confidentiality and prevent re-identification.